CLINICAL TRIAL: NCT02775110
Title: Natalizumab Temporary Discontinuation Study
Acronym: NaTDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, BNAC Director, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: USTYS0910017/JNI-2010-31
Record Dates: First submitted 2015-12-29; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Discontinuation Group (Active Comparator): Patients will discontinue the natalizumab therapy at once and initiate another disease modifying therapy at 1 month following the last natalizumab infusion. The disease modifying therapy at 1 month following natalizumab discontinuation will be at the discretion of the neurologist and may differ among patients.
  Interventions: Other: Natalizumab discontinuation
- Taper-off Group (Experimental): Patients will be administered two more natalizumab infusion, one at six weeks and the second at eight weeks (14 weeks from study entry), followed by six months natalizumab discontinuation. Another DMT will be initiated within two months after the last natalizumab infusion.
  Interventions: Other: Natalizumab discontinuation

INTERVENTIONS:
Other: Natalizumab discontinuation — Patients will be randomized to one of two groups: The Immediate Discontinuation Group (stop natalizumab immediately and continue with new DMT 1 month afterward) and the Taper-off Group (two additional infusions of natalizumab, one at 6 weeks and the next at 8 weeks following discontinuation. A new DMT will be initiated within 2 months of final natalizumab infusion).

SUMMARY:
This study evaluates the discontinuation of natalizumab either immediately or tapered off in the treatment of multiple sclerosis. Half of the fifty (50) participants will discontinue natalizumab immediately and the other half will taper off the drug, having two additional infusions, one at six weeks- and one at eight weeks-post discontinuation.

DETAILED DESCRIPTION:
Natalizumab is a pharmaceutical intervention used in the management of multiple sclerosis.

The decision to discontinue natalizumab therapy is often raised in patients defined as high-risk for PML despite good clinical efficacy. During the therapy cessation period following large phase III trials, a return to the prestudy disease activity was reached by four months post-discontinuation. Shorter therapy was associated with a trend for a more severe disease activity pointing to a possible 'rebound' effect after natalizumab discontinuation.

This study focuses on two different approaches: an immediate versus a step-wise/tapered down natalizumab discontinuation protocol, both with reinstitution of a different disease modifying therapy (DMT) within 1-6 months from the last natalizumab infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsing-remitting or relapsing-progressive (relapsing-remitting with incomplete recovery and secondary progressive with superimposed relapses) MS according to the McDonald criteria who have been on natalizumab therapy for at least 12 months
* Age 18-65
* Have EDSS scores less than or equal to 7.0
* Positive John Cunningham (JC) virus antibody results at screening
* Signed informed consent
* None of the exclusion criteria

Exclusion Criteria:

* Patients not willing or able to personally provide informed consent (subjects with cognitive impairment that effects the ability to provide informed consent for participation)
* Patients with active disease per clinical and MRI evaluation at baseline
* Patients with renal disease that precludes having an MRI with gadolinium contrast

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of recorded infections including viral opportunistic infection | Up to 1 year follow-up
  Number of recorded infections including viral opportunistic infections (i.e., shingles) will be recorded up to 1-year follow-up; continuous close vigilance will be maintained for possible cases of progressive multifocal leukoencephalopathy (PML)
Saturation percentage of α4β1integrin receptors on the surface of lymphocytes | 12 months
Number gadolinium-enhancing lesions | Change between baseline-6 months, 6 months-12 months, and baseline-12 months
  Number of gadolinium-enhancing lesions
Absolute changes in gadolinium-enhancing and T2-weighted lesion volume between timepoints | Change between baseline-6 months, 6 months-12 months, and baseline-12 months
  Absolute changes in gadolinium-enhancing and T2-weighted lesion volume
Sum of new and enlarging T2-weighted lesions | Change between baseline-6 months, 6 months-12 months, and baseline-12 months
  Sum of new and enlarging lesions as seen on T2-weighted images

SECONDARY OUTCOMES:
Number of clinical relapses | Either baseline (immediate discontinuation group) or 6 months (taper-off group)
  Number of clinical relapses will be assessed at the time of natalizumab therapy discontinuation which will be different between the two groups
Expanded Disability Status Scale (EDSS) score | Either baseline (immediate discontinuation group) or 6 months (taper-off group)
  Expanded disability status scale score

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Weinstock-Guttman, MD, Principal Investigator — Jacob's Neurological Institute
Locations (2):
- United States (2):
  - Buffalo Neuroimaging Analysis Center, Buffalo, New York
  - Jacobs Neurological Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No